CLINICAL TRIAL: NCT05832346
Title: Preliminarily Effects of a Laughter Yoga Program on the Mood, Anxiety, and Loneliness Among Adolescents With Intellectual and Physical Disabilities in a Special School: a Pilot Randomized Controlled Trial
Brief Title: Effects of a Laughter Yoga Program in Adolescents With Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEE Regina Lai Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022.660-T
Record Dates: First submitted 2023-02-06; First posted 2023-04-27 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Disability, Adolescent Learning; Psychosocial Problem
Keywords: disabilities; adolescents; psychosocial problems; laughter yoga; feasibility studies; randomized controlled trial
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Participant
Masking Description: masking the participants that they do not know which group will be allocated in this pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga programme (Experimental): The intervention group will receive a 4-week laughter yoga programme (8 sessions). This group also receives routine care provided by the special school as usual.
  Interventions: Behavioral: Laughter yoga programme
- Routine care (No Intervention): The control group receives routine care provided by the special school as usual.

INTERVENTIONS:
Behavioral: Laughter yoga programme — Intervention for intervention group:
  This is a 4-week laughter yoga programme (8 sessions) to help adolescents with intellectual and physical disabilities bring more happiness, laughter and joy to promote their mental health status. As laughter yoga therapy can reduce people's levels of stress, anxiety, depression, loneliness, strengthen the immune system and keep the mind positive. Each laughter yoga session will last for 15 minutes and in total there will be 8 sessions for four weeks (two sessions per week). Each laughter yoga session consists of hand clapping warming-up exercise, followed by deep breathing exercise, childlike playfulness exercise, and then laughter exercise. The intervention group also receives routine care provided by special school.
  Arms: Laughter yoga programme

SUMMARY:
A pilot randomized controlled trial will be adopted. A total of forty adolescents with intellectual and physical disabilities will be randomly allocated into either intervention group receiving a 4-week laughter yoga programme (8 sessions) or control group receiving routine care in a 1:1 ratio based on computer-generated random schedule. The aim of this pilot study is to preliminarily evaluate the effects of a 4-week laughter yoga programme (8 sessions) on the mood, anxiety and loneliness among adolescents with intellectual and physical disabilities in a special school in Hong Kong.

Hypotheses for primary outcomes of this study are as follows:

H.1 Participants receiving the 4-week laughter yoga programme (8 sessions) (intervention group) will have a greater improvement on mood level than the participants receiving routine care provided by the special school as usual (control group).

H.2 Participants receiving the 4-week laughter yoga programme (8 sessions) (intervention group) will have a greater reduction on anxiety than the participants receiving routine care provided by the special school as usual (control group).

H.3 Participants receiving the 4-week laughter yoga programme (8 sessions) (intervention group) will have a greater reduction on loneliness than the participants receiving routine care provided by the special school as usual (control group).

DETAILED DESCRIPTION:
Intervention

The purpose of a 4-week laughter yoga programme (8 sessions) combined with mindfulness activities is to help adolescents with intellectual and physical disabilities bring more happiness, laughter and joy to promote their mental health status. As the laughter yoga programme can reduce people's levels of stress, anxiety, loneliness and strengthen the immune system and keep the mind positive.

The elements in the protocol for implementing 15 minutes laughter yoga per session is adopted from the International Laughter Yoga for children with special needs:

1. Begins the first exercise: laughing solidly for five minutes with the following body and hands movements. You should keep moving your body.
2. Starts pulling faces: trying to emphasize your laughter- everyone should copy and follow.
3. Do hand gestures while laughing: Flick both hands and try to shark water off both hands.
4. Then apply invisible sun cream to your face.
5. Move the body to right and left with both hands up Five minutes pass and the participants should feel exhausted. Then, repeated same steps for two more times with a total of 15 minutes per session each day.

Study participants

The adolescents aged 10-18 years old with intellectual and physical disabilities will be recruited from a special school in Hong Kong. This special school locates in Diamond Hill in Kowloon side of Hong Kong and it is a medium size special school enrolls from mild to moderate students with intellectual and physical disabilities. Forty adolescents with mild to moderate physical and intellectual disabilities (ID) will be randomly allocated to either intervention group or control by the research team with a concealed envelop in a ratio of 1:1.

Study instruments

There are four sessions in this questionnaire including the demographic sheet, Mood Scale, State-Trait Anxiety Inventory (STAI-6), and Loneliness Scale for adolescents.

Data Collection

A briefing session will be delivered to the direct care staff in the school, school nurses and schoolteachers who will assist the participants to complete the questionnaire and demographic sheet with their understanding and behavioural observations.

The data collection will be conducted in both groups before and immediately after the intervention. Pre-test data collection will be conducted one week prior to the intervention. Post-test data collection will be conducted immediately after the intervention for both intervention and control groups.

Data analysis

Appropriate descriptive statistics, such as mean (standard deviation), median (inter-quartile range) and frequency (percentage) will be used to summarize and present the baseline characteristics and outcome data of the participants. Normality of continuous variables will be assessed based on their skewness and kurtosis statistics, values within ±2 indicating the plausibility of normal distribution. Suitable transformations will be made on skewed variables before subjecting them into inferential analysis. Homogeneity of baseline characteristics between the intervention and control groups will be assessed using independent t, chi-square or Fisher's exact tests, as appropriate. Multiple regression will be used to compare the change of each outcome at post-test with respect to pre-test between the two groups with adjustment for the pre-test level. All statistical analyses will be performed using IBM SPSS with level of significance set at 0.05 (2-sided).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent has been diagnosed with mild and moderate intellectual or/and physical disabilities
* Adolescent is studying between Grade 4 and Grade 12 in the selected special school
* Adolescent aged between 10 and 19 years old in this selected special school during the data collection period
* Adolescent has not received any psychotherapy previously
* Adolescent has the proficiency in understanding instructions for laughter exercises and hands and body movement

Exclusion Criteria:

* Adolescent has not been diagnosed with mild and moderate intellectual or/and physical disabilities
* Adolescent is studying lower than Grade 4 in the selected special school
* Adolescent aged < 10 years old and > 19 years old in this selected special school during the data collection period
* Adolescent has previously received psychotherapy
* Adolescent does not have the proficiency in understanding instructions for laughter exercises and hands and body movement

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Mood | Before the intervention
  The Mood Scale includes five different emoji with a 5-points response scale of mood ranging from 1-5: 1-Very bad; 2-bad, 3-so-so, 4-good; to 5-very good. The range of scale score can be from 1 to 5 where higher scores represented very good mood and emotion using emoji.
Mood | Immediate after the intervention
  The Mood Scale includes five different emoji with a 5-points response scale of mood ranging from 1-5: 1-Very bad; 2-bad, 3-so-so, 4-good; to 5-very good. The range of scale score can be from 1 to 5 where higher scores represented very good mood and emotion using emoji.
Anxiety | Before the intervention
  The STAI-6 contains 6 items which is sensitive to fluctuations in state anxiety. Observers will be asked to answer each item using the following scale (Scale of 1-5; 1 = not at all / very slightly, 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely). The range of score from 6 to 24. The highest score shows a high anxiety level of individual. Back translation of the STAI-6 had been performed after obtained the content validity index (CVI=1.0).
Anxiety | Immediate after the intervention
  The STAI-6 contains 6 items which is sensitive to fluctuations in state anxiety. Observers will be asked to answer each item using the following scale (Scale of 1-5; 1 = not at all / very slightly, 2 = a little, 3 = moderately, 4 = quite a bit, 5 = extremely). The range of score from 6 to 24. The highest score shows a high anxiety level of individual. Back translation of the STAI-6 had been performed after obtained the content validity index (CVI=1.0).
Loneliness | Before the intervention
  The UCLA Loneliness Scale (ULS-8) contains 8 items including two factors: intimate other and social other. There are six items in the intimate factor and two items in the social other factor. Observers are asked to answer each item using the following scale: 1=Never, 2=Rarely, 3=Sometimes, 4=Often. It is a 4-point Likert scale with values from "never" to "always". For each participant, responses on the 4-items were totaled to create a composite loneliness score, with higher scores indicated higher loneliness. Scores ranged from 8 to 32. The 8-item measure demonstrated high internal reliability (α=0.84).
Loneliness | Immediate after the intervention
  The UCLA Loneliness Scale (ULS-8) contains 8 items including two factors: intimate other and social other. There are six items in the intimate factor and two items in the social other factor. Observers are asked to answer each item using the following scale: 1=Never, 2=Rarely, 3=Sometimes, 4=Often. It is a 4-point Likert scale with values from "never" to "always". For each participant, responses on the 4-items were totaled to create a composite loneliness score, with higher scores indicated higher loneliness. Scores ranged from 8 to 32. The 8-item measure demonstrated high internal reliability (α=0.84).

CONTACTS AND LOCATIONS:
Overall Officials: Regina Lee, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Nethersole School of Nursing, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
It is anonymous data and it will be shared upon request.
Supporting Information: Study Protocol
Time Frame: In 6 months after the submission of the final report.
Access Criteria: Once the personal data management account has been set up.

REFERENCES:
- [Background] Hall, L.; Hume, C.; Tazzyman, S. Five degrees of happiness: Effective Smiley Face Likert Scales for evaluating with children. In Proceedings of the 15th International Conference on Interaction Design and Children, Manchester, UK, 21-24 June 2016; pp. 311-321. https://dl.acm.org/doi/proceedings/10.1145/2930674
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Wilson D, Cutts J, Lees I, Mapungwana S, Maunganidze L. Psychometric properties of the revised UCLA Loneliness Scale and two short-form measures of loneliness in Zimbabwe. J Pers Assess. 1992 Aug;59(1):72-81. doi: 10.1207/s15327752jpa5901_7. PMID 1512681